CLINICAL TRIAL: NCT04542122
Title: Moral Judgements and Choices of Caregivers in the Time of COVID-19 Pandemic: a Randomized Experimental Study
Brief Title: Moral Judgements and Choices of Caregivers in the Time of COVID-19 Pandemic
Acronym: XPHI-COVID19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 1474
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-07

CONDITIONS: Morals
Keywords: morals; ethics; moral judgements; moral choices; covid 19; survey; utilitarianism; deontology; oxford utilitarianism scale
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choices then judgements (No Intervention)
- Judgements then choices (Active Comparator): Switch in the order of clinical cases in the survey
  Interventions: Behavioral: Choices and judgements

INTERVENTIONS:
Behavioral: Choices and judgements — In the intervention arm, the participant is asked to answer clinical cases in a reverse order from the control group (control has to make moral choices then judge somebody else's choices ; intervention has to judge moral choices first, then make his own)
  Arms: Judgements then choices

SUMMARY:
The XPHI-COVID19 randomized study aims to investigate the mechanisms of moral judgements in a population of caregivers, using a survey, with the results to the Oxford Utilitarianism Scale as primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* All caregivers from french public healthcare center with Intensive Care Unit
* Agreement

Exclusion Criteria:

* Refuse to participate or withdraw agreement

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-09-03 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-08-02 (Estimated)

PRIMARY OUTCOMES:
Oxford Utilitarianism Scale | Up to one year
  Two-Dimensional Model of Utilitarian Psychology

CONTACTS AND LOCATIONS:
Overall Officials: Clement GAKUBA, MD PhD, Principal Investigator — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahane G, Everett JAC, Earp BD, Caviola L, Faber NS, Crockett MJ, Savulescu J. Beyond sacrificial harm: A two-dimensional model of utilitarian psychology. Psychol Rev. 2018 Mar;125(2):131-164. doi: 10.1037/rev0000093. Epub 2017 Dec 21. PMID 29265854
- [Background] Garbutt G, Davies P. Should the practice of medicine be a deontological or utilitarian enterprise? J Med Ethics. 2011 May;37(5):267-70. doi: 10.1136/jme.2010.036111. Epub 2011 Jan 29. PMID 21278402
- [Background] Conway P, Goldstein-Greenwood J, Polacek D, Greene JD. Sacrificial utilitarian judgments do reflect concern for the greater good: Clarification via process dissociation and the judgments of philosophers. Cognition. 2018 Oct;179:241-265. doi: 10.1016/j.cognition.2018.04.018. Epub 2018 Jul 2. PMID 30064654
- [Background] Einav S, Benoit DD. Focus on ethics of admission and discharge policies and conflicts of interest. Intensive Care Med. 2019 Aug;45(8):1130-1132. doi: 10.1007/s00134-019-05673-3. Epub 2019 Jul 2. No abstract available. PMID 31267194
- [Background] Emanuel EJ, Persad G, Upshur R, Thome B, Parker M, Glickman A, Zhang C, Boyle C, Smith M, Phillips JP. Fair Allocation of Scarce Medical Resources in the Time of Covid-19. N Engl J Med. 2020 May 21;382(21):2049-2055. doi: 10.1056/NEJMsb2005114. Epub 2020 Mar 23. No abstract available. PMID 32202722
- [Background] Truog RD, Mitchell C, Daley GQ. The Toughest Triage - Allocating Ventilators in a Pandemic. N Engl J Med. 2020 May 21;382(21):1973-1975. doi: 10.1056/NEJMp2005689. Epub 2020 Mar 23. No abstract available. PMID 32202721
- [Background] Leclerc T, Donat N, Donat A, Pasquier P, Libert N, Schaeffer E, D'Aranda E, Cotte J, Fontaine B, Perrigault PF, Michel F, Muller L, Meaudre E, Veber B. Prioritisation of ICU treatments for critically ill patients in a COVID-19 pandemic with scarce resources. Anaesth Crit Care Pain Med. 2020 Jun;39(3):333-339. doi: 10.1016/j.accpm.2020.05.008. Epub 2020 May 17. PMID 32426441
- [Background] Rosenbaum L. Facing Covid-19 in Italy - Ethics, Logistics, and Therapeutics on the Epidemic's Front Line. N Engl J Med. 2020 May 14;382(20):1873-1875. doi: 10.1056/NEJMp2005492. Epub 2020 Mar 18. No abstract available. PMID 32187459